CLINICAL TRIAL: NCT06149169
Title: An Open-Label, Single-Arm Study of Relma-cel, CD19-targeted Chimeric Antigen Receptor (CAR)T Cells for Relapsed and Refractory (R/R) LBCL
Brief Title: CD19-targeted CAR T Cells for Relapsed and Refractory (R/R) Large B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029-017
Record Dates: First submitted 2023-11-14; First posted 2023-11-28 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-03

CONDITIONS: Lymphoma, Non-Hodgkin; Diffuse Large B Cell Lymphoma
Keywords: JWCAR029; B-Cell Malignancies; CAR T cells; Chimeric antigen receptor; Relapsed/Refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relma-cel (Experimental): The PK, safety and efficacy of Relma-cel will be evaluated in 1 x 10^8 CAR+T cells dose level
  Interventions: Biological: CD19-targeted Chimeric Antigen Receptor(CAR) T Cells

INTERVENTIONS:
Biological: CD19-targeted Chimeric Antigen Receptor(CAR) T Cells — Relma-cel be administered at one dose level:1×10^8 CAR+T cells

SUMMARY:
This is an open-label, single-arm study to treat the adult R/R Large B-cell Lymphoma subjects with Relmacabtagene autoleucel (relma-cel) in China.

DETAILED DESCRIPTION:
This is an open-label, single-arm study conducted in adult subjects with R/R LBCL in China to evaluate the pharmacokinetics(PK), safety and efficacy of relma-cel, monitor the immune response after relma-cel treatment.

Relma-cel was approved by the China National Medical Products Administration(NMPA)in September 2021(Acceptance No:CXSS2000036)for the treatment of adult patients with R/R LBCL after second-line or more systemic therapy.The recommended dose is 1×10^8 CAR+T cells.The indication for this application is R/R LBCL(supplement study) and the recommended dose is 1×10^8 CAR+T cells.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. Sign on the informed consent;
3. Subjects must have histologically confirmed Large B-cell Lymphoma;
4. Subjects had been treated with anthracyclines and rituximab(or other CD20-targeted antibodies) and had relapsed, failed to respond, or progressed after at least two lines of therapy include autologous hematopoietic stem cell transplantation(auto-HSCT);
5. Subjects have accessible PET-positive lesion and have measurable CT-positive lesion according to Lugano Classification;
6. Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1;
7. Adequate organ function;
8. Adequate vascular access for leukapheresis procedur;
9. Subjects who have previously received CD19 targeted therapy must confirm that lymphoma lesions still expresss CD19;
10. Women of childbearing potential must agree to use highly effective methods of contraception for 1 year after the last dose of Relma-cel;
11. Males who have partners of childbearing potential must agree to use an effective barrier contraceptive method for 1 year after the last dose of Relma-cel.

Exclusion Criteria:

1. Central nervous system(CNS) only involvement by malignancy or primary CNS lymphoma;
2. History of another primary malignancyn that has not been in remission for at least 2 years;
3. Subjects has HBV,HCV,HIV or syphilis nefection at the time of screening;
4. Active deep venous thrombosis(DVT)/Pulmonary embolism(PE),or active DVT/PE requires anti-coagulation within 3 months prior to signing the ICF;
5. Subjects with uncontrolled systemic fungal,bacterial,viral or other infection;
6. Presence of acute or chronic graft-versus-host disease(GVHD);
7. History of any serious cardiovascular disease or presence of clinically relevant CNS pathology;
8. Pregnant or nursing woman;
9. Subjects using of any chemotherapy,corticisteriod,experiment agents,GVHD therapies,radiation,allo-HSCT or any other therapies for lymphoma must go through a specific wash-out period before leukapheresis;
10. Uncontrolled conditions or unwillingness or inability to follow the procedures required in the protocol;
11. Received CAR T-cell or other genetically-modified T-cell therapy previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic(PK)-Cmax of Relma-cel | up to 1 year after Relma-cel infusion
  Maximum observed concentration of Relma-cel in peripheral blood
Pharmacokinetic(PK)-Tmax of Relma-cel | up to 1 year after Relma-cel infusion
  Time to maximum concentration of Relma-cel in peripheral blood
Pharmacokinetic(PK)-AUC of Relma-cel | up to 1 year after Relma-cel infusion
  Area under the concentration vs time curve of Relma-cel

SECONDARY OUTCOMES:
Objective response rate (ORR) in LBCL subjects | 3 months
  Objective response rate (ORR) in 3 month evaluated by investigator of LBCL subjects.
Best objective response rate ( Best ORR) in LBCL subjects | up to 1 year after Relma-cel infusion
  Best objective response rate (ORR) evaluated by the investigator of LBCL subjects.
Complete response rate (CRR) in LBCL subjects | up to 1 year after Relma-cel infusion
  Complete response rate (CRR) at any time points evaluated by the investigator.
Adverse events (AEs) | up to 1 year after Relma-cel infusion
  These adverse events would be measured by assessment scale method according to NCI-CTCAE v4.03 classification standard.
Duration of response (DOR) | up to 1 year after Relma-cel infusion
  Time from first response (PR or CR) to disease progression or death from any cause.
Progression-free survival (PFS) | up to 1 year after Relma-cel infusion
  Progression-free survival
Overall survival (OS) | up to 1 year after Relma-cel infusion
  Overall survival
Changes of serum cytokines-IL-2，IL-6，IL-8 and IFN- γ | up to 1 year after Relma-cel infusion
  The changes of serum cytokines-IL-2，IL-6，IL-8 and IFN- γ after Relma-cel infusion.
Changes of inflammation biomarker-CRP | up to 1 year after Relma-cel infusion
  The changes of inflammation biomarker-CRP after Relma-cel infusion.
Changes of inflammation biomarker-serum ferritin | up to 1 year after Relma-cel infusion
  The changes of inflammation biomarker-serum ferritin after Relma-cel infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Huilai Zhang, Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No